CLINICAL TRIAL: NCT02065011
Title: An Open-label Study to Determine the Long-term Safety, Tolerability and Biological Activity of SAR421869 in Patients With Usher Syndrome Type 1B
Brief Title: A Study to Determine the Long-Term Safety, Tolerability and Biological Activity of SAR421869 in Patients With Usher Syndrome Type 1B
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LTS13619; 2024-513500-34 (Registry Identifier: CTIS); US1/002/13 (Other: Sanofi Identifier); 2013-000597-29 (EudraCT Number)
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Usher's Syndrome
MeSH Terms: conditions — Usher Syndromes | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Long-term follow up (Other): Long-term follow up of patients who received SAR421869 in a previous study TDU13600
  Interventions: Drug: Blood draw for the laboratory assessment

INTERVENTIONS:
Drug: Blood draw for the laboratory assessment

SUMMARY:
Primary Objective:

To evaluate the long-term safety and tolerability of SAR421869 in patients with Usher syndrome Type 1B

Secondary Objective:

To assess long-term safety and biological activity of SAR421869

DETAILED DESCRIPTION:
The total duration of study period is up to 15 years.

ELIGIBILITY:
Inclusion criteria :

Provide signed and dated written informed consent (and if appropriate assent) and any locally required authorization eg, Health Insurance Portability and Accountability Act (HIPAA).

Must have been enrolled in protocol TDU13600. Must have received a subretinal injection of SAR421869

Exclusion criteria:

Did not receive SAR421869 as part of the TDU13600 protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-09-12 (Actual); Primary Completion 2031-06-13 (Estimated); Study Completion 2031-06-13 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events | 15 years
  The number and percentage of patients with treatment emergent adverse events

SECONDARY OUTCOMES:
Clinically important changes in ocular safety assessments | baseline to 15 years
  From baseline in (TDU13600) study and from the last visit best-corrected visual acuity (BCVA), slit-lamp examination, fundososcopy, intraocular pressure, laboratory parameters, concomitant medications
Delay in retinal degeneration | baseline to 15 years
  Measured as change from baseline in function relative to untreated contralateral eye on: BCVA, static perimetry, autofluorescence, optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, MD, Study Director — Sanofi
Locations (2):
- Oregon Health and Science University Site Number : 840001, Portland, Oregon, United States
- Investigational Site Number : 250001, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LTS13619 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26098&tenant=MT_SNY_9011